CLINICAL TRIAL: NCT05034146
Title: The Diagnostic Efficiency of 68Ga-FAPI PET/CT in Malignant Tumors
Brief Title: 68Ga-FAPI PET/CT in Malignant Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Principal Investigator, Yong He, principal investigator, Zhongnan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ZNYYHYXK0001
Record Dates: First submitted 2021-08-25; First posted 2021-09-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Fibroblast Activation Protein Inhibitor; PET/CT; Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — 68Ga-FAPI; Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Intervention Model Description: Experimental: 68Ga-FAPI PET/CT Investigators select subjects from patients who have underwent whole-body 18F-FDG PET/CT scan for suspected or confirmed malignancy, or suspected recurrence and metastasis after treatment for malignant tumors, focusing on malignant tumors with low FDG uptake including glioma, hepatocellular carcinoma, renal cancer, gastrointestinal cancer, and peritoneal metastases. Then the subjects receive whole-body 68Ga-FAPI PET/CT scan with time interval of one to four week.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 68Ga-FAPI PET/CT in malignant tumors (Experimental): Investigators select subjects from patients who have underwent whole-body 18F-FDG PET/CT scan for suspected or confirmed malignancy, or suspected recurrence and metastasis after treatment for malignant tumors, focusing on malignant tumors with low FDG uptake including glioma, hepatocellular carcinoma, renal cancer, gastrointestinal cancer, and peritoneal metastases. Then the subjects receive whole-body 68Ga-FAPI PET/CT scan with time interval of one to four week.
  Interventions: Drug: 68Ga-FAPI; Device: PET/CT

INTERVENTIONS:
Drug: 68Ga-FAPI — 68Ga-FAPI was injected intravenously to each subject, and the dose is calculated according to body weight of subject (approximately 1.85-3.7MBq/kg).
  Other Names: 68Ga-fibroblast activation protein inhibitor
Device: PET/CT — 68Ga-FAPI PET/CT scan were performed 20~60 min after 68Ga-FAPI (1.85-3.7MBq/kg) injection intravenously.
  Other Names: positron emission tomography/computed tomography

SUMMARY:
Fibroblast-activation protein (FAP) is a type Ⅱ transmembrane serine protease and is overexpressed in cancer-associated fibroblasts (CAFs). CAFs are the predominant component in the stroma of epithelial neoplasms. FAP can be detected in various of malignant neoplasms and is associated to tumor cell migration, invasion, and angiogenesis. Recently, a novel molecular probe, gallium 68-labelled FAP inhibitor (68Ga-FAPI), has been developed and used for visualization of tumor stroma by targeting FAP. Recent studies show favorable diagnosis efficiency in a variety of tumors, especially in gastrointestinal cancer, but the previous studies were all small-sample data or case reports. Therefore, further large-size research is necessary to confirm the advantages of 68Ga-FAPI in various of malignant tumors.

DETAILED DESCRIPTION:
The morbidity and mortality of malignant tumors are increasing. It is one of the major diseases that affect human health. At present, the conventional imaging diagnosis methods of a variety of malignant tumors are mainly CT and MRI based on anatomical imaging. Different from traditional imaging methods to visually display the lesion, nuclear medicine molecular imaging can not only locate the tumor location, but also image the expression and activity of specific molecules and biological processes. This molecular imaging method integrating anatomy and function is a noninvasive imaging to realize the early diagnosis and differential diagnosis, curative effect evaluation and follow-up observation of a variety of tumors. Positron emission tomography/computed tomography (PET/CT) uses specific molecular probes to target tumor. It can provide detailed information about the biochemical changes of tumor tissues at the cellular and molecular levels. It has better sensitivity and specificity than conventional imaging methods. At present, the most commonly used imaging agent in clinic is 18F-fluorodeoxyglucose (18F-FDG). 18F-FDG PET/CT is a valuable imaging modality in the management of patients with malignant tumors, but it is not a specific imaging agent for tumor application. The physiological uptake of gastrointestinal tract, infected tissues, or inflammatory cells can cause high 18F-FDG uptake resulting in a significant increase of the false positive rate; in addition, some tumors including well-differentiated hepatocellular carcinoma, renal cell carcinoma, and gastric signet ring cell carcinoma have low 18F-FDG uptake resulting in a high false negative rate. Therefore, it is very important to develop new molecular probes for targeting tumor.

Fibroblast-activation protein (FAP) is a type Ⅱ transmembrane serine protease and is overexpressed in cancer-associated fibroblasts (CAFs). CAFs are the predominant component in the stroma of epithelial neoplasms. FAP can be detected in various of malignant neoplasms and is associated to tumor cell migration, invasion, and angiogenesis. Recently, a novel molecular probe, gallium 68-labelled FAP inhibitor (68Ga-FAPI), has been developed and used for visualization of tumor stroma by targeting FAP. Recent studies show favorable diagnosis efficiency in a variety of tumors, especially in gastrointestinal cancer, but the previous studies were all small-sample data or case reports. Therefore, further large-size research is necessary to confirm the advantages of 68Ga-FAPI in various of malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

Volunteering to participate in clinical trial and sign an informed consent form Patients with suspected or confirmed malignant tumor

Exclusion Criteria:

Female patients plan to become pregnant within 6 months Pregnant and lactating women Patients are allergic to multiple drugs including test drug Patients have participated in other clinical trials in the past one month

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-02-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The diagnostic sensitivity and specificity of 68Ga-FAPI PET/CT in the staging of malignant tumors | three years
  Taking the pathology or clinical follow-up as gold standard, the sensitivity and specificity of 68Ga-FAPI PET/CT in detecting malignant tumor were calculated.

SECONDARY OUTCOMES:
Prognostic value of FAPI PET parameters in malignant tumors | From baseline to 1 year post-treatment
  Correlation between FAPI PET parameters (SUVmax/SUVmean/SUVpeak, measured in the Syngo Workstation (Siemens Healthineers)) and long-term outcomes (e.g., progression-free survival, overall survival).
FAPI PET for therapeutic response evaluation in malignant tumors | Within 1 week after completion of neoadjuvant or adjuvant therapy
  Assessment of FAPI PET parameters, namely SUVmax, SUVmean, SUVpeak, measured in the Syngo Workstation (Siemens Healthineers), for evaluating treatment response in patients with malignant tumors.
The connection between FAPI PET parameters and histopathological biomarkers. | Within 4 weeks of FAPI PET scan
  Analyze the correlation between FAPI PET parameters (SUVmax/SUVmean/SUVpeak, measured in the Syngo Workstation (Siemens Healthineers)) and FAP expression levels (H-score; immunohistochemistry) or immune - related biomarkers, such as PD-L1 expression (Combined Positive Score; Dako 22C3 IHC assay), CD8 expression (H-score; immunohistochemistry), Granzyme B expression (H-score; immunohistochemistry).

CONTACTS AND LOCATIONS:
Overall Officials: Yong He, MD, PhD, Principal Investigator — Zhongnan Hospital
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kratochwil C, Flechsig P, Lindner T, Abderrahim L, Altmann A, Mier W, Adeberg S, Rathke H, Rohrich M, Winter H, Plinkert PK, Marme F, Lang M, Kauczor HU, Jager D, Debus J, Haberkorn U, Giesel FL. 68Ga-FAPI PET/CT: Tracer Uptake in 28 Different Kinds of Cancer. J Nucl Med. 2019 Jun;60(6):801-805. doi: 10.2967/jnumed.119.227967. Epub 2019 Apr 6. PMID 30954939
- [Background] Pang Y, Zhao L, Luo Z, Hao B, Wu H, Lin Q, Sun L, Chen H. Comparison of 68Ga-FAPI and 18F-FDG Uptake in Gastric, Duodenal, and Colorectal Cancers. Radiology. 2021 Feb;298(2):393-402. doi: 10.1148/radiol.2020203275. Epub 2020 Dec 1. PMID 33258746
- [Derived] Li H, Li C, Tian Y, Xiao Z, Xing D, He Y. Same-day dual-tracer PET/CT imaging with [68 Ga]Ga-FAPI-04 following [18F]FDG finds answers in patients presenting with negative or equivocal [18F]FDG. Ann Nucl Med. 2025 Nov;39(11):1237-1248. doi: 10.1007/s12149-025-02080-1. Epub 2025 Jul 4. PMID 40614035
- [Derived] Jiang Y, Yu Z, Sun Y, Tian Y, Wang L, Xing D, Huang Y, He Y, Jia J. Predictive value of [68Ga]Ga-FAPI-04 PET/CT on pathologic response to neoadjuvant chemoimmunotherapy for locally advanced resectable oral squamous cell carcinoma. Eur J Nucl Med Mol Imaging. 2025 Dec;53(1):283-294. doi: 10.1007/s00259-025-07414-9. Epub 2025 Jun 23. PMID 40548990
- [Derived] Jiang Y, Huang S, Tian Y, Xing D, Xiao Z, Huang J, He Y. Dual-Time Point 68 Ga-FAPI-04 PET/CT Improves Tumor Delineation and Cervical Lymph Node Metastasis Identification in Patients With Head and Neck Squamous Cell Carcinoma. Clin Nucl Med. 2025 Mar 1;50(3):e130-e137. doi: 10.1097/RLU.0000000000005610. Epub 2024 Dec 13. PMID 39668486
- [Derived] Chen J, Xu K, Li C, Tian Y, Li L, Wen B, He C, Cai H, He Y. [68Ga]Ga-FAPI-04 PET/CT in the evaluation of epithelial ovarian cancer: comparison with [18F]F-FDG PET/CT. Eur J Nucl Med Mol Imaging. 2023 Nov;50(13):4064-4076. doi: 10.1007/s00259-023-06369-z. Epub 2023 Aug 1. PMID 37526694